CLINICAL TRIAL: NCT07364539
Title: Local Registry of Central Nervous System Infections (ReCeNSI)
Acronym: ReCeNSI
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Raffaella Lissandrin, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: ReCeNSI
Record Dates: First submitted 2025-12-19; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-09

CONDITIONS: Central Nervous System (CNS) Infection
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
Central Nervous System (CNS) infections are considered rare conditions but at the same time, they are emergencies whose diagnosis and treatment are time-dependent. They include several clinical syndromes, including meningitis, encephalitis, brain abscesses, and post-surgical meningitis. The classic triad of symptoms includes fever, altered mental status, and neck stiffness, but other common manifestations include nausea and vomiting, cranial nerve dysfunction, skin rash, and seizures. Due to the potentially life-threatening effects on patients, these clinical conditions cannot be underestimated. The CNS includes the brain and spinal cord, surrounded and protected by the meninges and cerebrospinal fluid (CSF). Within the CNS are numerous nuclei responsible for vital functions, as well as more complex intellectual activities.

ELIGIBILITY:
* Pazients admitted to the Fondazione IRCSS Policlinico San Matteo
* Diagnosis of bacterial meningitis, meningoencephalitis, bacterial CNS infection, viral CNS infection, viral encephalitis, brain abscess, or post-neurosurgical meningitis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: In the nine years since 2012, we have identified 260 patients with positive CSF tests. We assume that over the next 10 years we will register the same number of patients, for a total of 520 patients. With this sample size, the precision of the mortality estimate over the study period will be at worst ±4.3%, corresponding to half the 95% confidence interval (CI) of a 50% chance. If the mortality rate were 10%, the precision would be ±2.7%; if the mortality rate were 5%, the precision would be ±2%.
Sampling Method: Non-Probability Sample
Enrollment: 520 (Estimated)
Dates: Start 2022-03-04 (Actual); Primary Completion 2022-03-05 (Actual); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the outcome in terms of mortality at discharge in patients with CNS infections. | From January 2012

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia, Italia, Italy